CLINICAL TRIAL: NCT00999349
Title: Combined Therapy of Silymarin and Desferrioxamine in Patients With B-thalassemia Major: a Randomized Double-blind Clinical Trial
Brief Title: Therapeutic Effects of Silymarin in Patients With B-thalassemia Major
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Madaus Inc (Industry)
Responsible Party: Professor Behjat Moayedi, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 187050; LE13K0.52,; IRCT138804022067N1
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Beta-thalassemia Major; Iron Overload
Keywords: iron overload condition; regular desferrioxamine administration; receiving continuous blood transfusions
MeSH Terms: conditions — beta-Thalassemia; Iron Overload | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Silymarin (LEGALON) (Experimental)
  Interventions: Drug: Silymarin (LEGALON)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silymarin (LEGALON) — Study group: Silymarin Capsule, 140 mg, 3 times a day + desferrioxamine injection 50 mg/kg, Placebo group:Placebo capsules Similar to Silymarin +desferrioxamine injection 50 mg/kg
  Arms: Silymarin (LEGALON)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Silymarin, a flavonolignan complex isolated from Silybum marianum, has a strong antioxidant, hepatoprotective and iron chelating activities. The present study has been designed to investigate the therapeutic activity of orally administered silymarin in patients with thalassemia major under conventional iron chelation therapy. A 6-month randomized, double-blind, clinical trial was conducted in 140 beta-thalassemia major patients in two well-matched groups. Patients are randomized to receive a silymarin tablet (140 mg) three times a day plus conventional desferrioxamine therapy or the same therapy but a placebo tablet instead of silymarin. Clinical laboratory tests of iron status and liver function are assessed at the beginning and the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Presence of major Beta-thalassemia
* Age 12 years or older
* Iron overload condition (serum ferritin levels between 1000-5000 ng/mL) Regular desferrioxamine administration (50 mg/kg)
* Continuous blood transfusions
* Negative CRP test

Exclusion criteria:

* Hepatitis B or C infection
* Positive HIV test
* Chronic renal or heart failure
* Iron chelating therapy with other iron chelators

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin level | after 3 months and 6 months from beginning of the trial

SECONDARY OUTCOMES:
Liver enzymes (SGOT, SGPT, Alkaline Phosphatase), serum Hepcidin, and soluble transferrin receptor levels | At the beginning and the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Behjat Moayedi, Professor, Principal Investigator — Isfahan University of Medical Sciences, moayedi@med.mui.ac.ir
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

REFERENCES:
- [Background] Gharagozloo M, Moayedi B, Zakerinia M, Hamidi M, Karimi M, Maracy M, Amirghofran Z. Combined therapy of silymarin and desferrioxamine in patients with beta-thalassemia major: a randomized double-blind clinical trial. Fundam Clin Pharmacol. 2009 Jun;23(3):359-65. doi: 10.1111/j.1472-8206.2009.00681.x. Epub 2009 May 7. PMID 19453758